CLINICAL TRIAL: NCT04412434
Title: EEG Patterns in Patients With Acute Ischemic Stroke Resulted From Large Vessels Occlusion in the Anterior Circulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: rambam62 (Other)
Responsible Party: Sponsor-Investigator, rambam62, Director, Head of Stroke Service, Principal Investigator, Clinical Professor, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0297-20 RMB
Record Dates: First submitted 2020-05-27; First posted 2020-06-02 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Stroke, Ischemic
Keywords: eeg pattern; acute ischemic stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients with acute ischemic stroke (Other): This open-label prospective study will be conducted in the single medical center (RAMBAM Medical Center) and will include at least 200 patients with acute ischemic stroke resulted from MCA or ICA occlusion.
  Interventions: Diagnostic Test: Electroencephalography (EEG)

INTERVENTIONS:
Diagnostic Test: Electroencephalography (EEG) — Electroencephalography (EEG) is a painless and harmless method to record the bioelectric activity of the brain. Clinically, EEG refers to the recording of the brain's spontaneous electrical activity over a period of time, as recorded from multiple electrodes placed on the scalp This method can be helpful in the diagnosis of many various brain diseases and pathological conditions.
  For the examination, electrodes are placed on the head, using a special harmless gel, similar to gel, used in ultrasonographic studies.

SUMMARY:
Clinical deterioration is observing in up to forty percent of patients with acute ischemic stroke (AIS) due to large vessels occlusion. Until now, there is no automated monitoring system for early detection of neurological deterioration in such patients. As a first step to develop such system investigators suggest this study aiming to evaluate patterns of brain electrical activity registered by EEG in patients with AIS attributed to the MCA or ICA territory correlated with location and extension of ischemic lesions as determined by non-contrast CT (NCT).

DETAILED DESCRIPTION:
Rationale. Despite the exciting developments in the treatment of acute ischemic stroke (AIS) in last years, the problem of neurological deterioration in patients with AIS remains unresolved and poorly understandable. This is especially correct about patients with AIS resulted from large vessel occlusion (LVO), mainly internal carotid artery (ICA) and middle cerebral artery (MCA) occlusion. Such deterioration is observing in up to forty percent of patients with acute ischemic stroke due to LVO. On the other side, according to the literature about 40 % of LVO strokes resulted from atrial fibrillation. Until now, there is no automated monitoring system for early detection of neurological deterioration in AIS patients. Such monitoring system may save millions of lives of stroke victims all over the world. As a first step to develop such system based on change of brain electrical activity registered by electroencephalography (EEG) in patients with AIS investigators suggest this study.

Overall goal. The aim of the suggested research is to evaluate patterns of brain electrical activity registered by EEG in patients with AIS attributed to the MCA or ICA territory in correlation with location and extension of ischemic lesions as determined by non-contrast CT (NCT). Based on these data, the attempt to find algorithms, describing such correlation will be done.

Target population. The prospective study will include at least 200 AIS patients with acute stroke resulted from MCA or ICA occlusion.

Methods. Non contrast CT and EEG will be done at the same day. Neurologist will evaluate neurological status at the day of EEG and CT performing and clinical score by National Institute of Health Stroke Scale (NIHSS) will be obtained. EEG will be performed continuously for at least 30 minutes with 19-channel EEG machine.

Assessment. After gathering clinical, EEG and NCT data mathematical and computerized analysis (including Artificial Intelligence methods) will be applied aiming to find algorithms describing relationship between size and location of AIS and change in brain electrical activity registered by EEG in AIS patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke, due to large vessel occlusion
* Age of 18 years and more
* Male or Female
* Modified Rankin Scale of ≤ 2 prior to presentation
* NIHSS ≥ 4 at the day of NCT and EEG

Exclusion Criteria:

* Epilepsy
* Brainstem or cerebellar stroke
* Intracranial or extracranial hemorrhage of any kind
* History of severe head trauma
* History of severe dementia or progressive neurodegenerative disease
* Cerebral tumor or hydrocephalus by anamnesis or by imaging
* Lacunar stroke
* Significant movement disorder.
* Local skull or skin condition, preventing EEG electrode application.
* Any known disorder, which may interfere with the protocol implementation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-04 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
EEG pattern | 24 months
  EEG patterns depending on size and location of acute ischemic stroke,including generalized or focal slowing or both and epileptiform discharges

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Telman, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam MC, Haifa, Israel